CLINICAL TRIAL: NCT00006379
Title: Purine-Analog-Containing Non-Myeloablative Allogeneic Stem Cell Transplantation for Treatment of Hematologic Malignancies and Severe Aplastic Anemia
Brief Title: Non-Ablative Allo HSCT For Hematologic Malignancies or SAA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU3Y00; P30CA043703 (NIH); CWRU-3Y00 (Other: Case Comprehensive Cancer Center); 05-00-07 (Other: University Hospitals IRB); NCI-G00-1868
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases; Precancerous/Nonmalignant Condition; Small Intestine Cancer
Keywords: monoclonal gammopathy of undetermined significance; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; small intestine lymphoma; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; polycythemia vera; chronic idiopathic myelofibrosis; essential thrombocythemia; adult acute erythroid leukemia (M6); adult acute megakaryoblastic leukemia (M7); childhood acute erythroleukemia (M6); childhood acute megakaryocytic leukemia (M7); recurrent/refractory childhood Hodgkin lymphoma; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; acute undifferentiated leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; prolymphocytic leukemia; primary systemic amyloidosis; adult acute minimally differentiated myeloid leukemia (M0); childhood acute minimally differentiated myeloid leukemia (M0); recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; childhood chronic myelogenous leukemia; chronic eosinophilic leukemia; chronic neutrophilic leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; juvenile myelomonocytic leukemia; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12); childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Precancerous Conditions; Monoclonal Gammopathy of Undetermined Significance; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Recurrence; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Mycosis Fungoides; Sezary Syndrome; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myelomonocytic, Juvenile; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Congenital Abnormalities | interventions — Antilymphocyte Serum; Cyclophosphamide; fludarabine phosphate; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: anti-thymocyte globulin — anti-thymocyte globulin IV over at least 4 hours on days -2 and -1
Biological: graft-versus-tumor induction therapy — Patients undergo filgrastim (G-CSF)-mobilized allogeneic peripheral blood stem cell transplantation on day 0.
Drug: cyclophosphamide — cyclophosphamide IV over 2 hours on days -3 to -2
Drug: fludarabine phosphate — fludarabine IV over 30 minutes on days -8 to -4
Procedure: peripheral blood stem cell transplantation — Patients undergo filgrastim (G-CSF)-mobilized allogeneic peripheral blood stem cell transplantation on day 0.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy used to kill cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by peripheral stem cell transplantation in treating patients who have hematologic cancer or aplastic anemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the rates of durable full donor hematologic engraftment in patients with high-risk hematologic malignancies or severe aplastic anemia treated with non-myeloablative conditioning using fludarabine, cyclophosphamide, and anti-thymocyte globulin followed by allogeneic peripheral blood stem cell transplantation.
* Determine the acute and delayed toxic effects of this non-myeloablative conditioning regimen in this patient population.
* Determine the event-free and overall survival of patients treated with this regimen.
* Determine the incidence and severity of acute and chronic graft-versus-host disease in patients treated with this regimen.
* Determine the rate and quality of immune reconstitution in patients treated with this regimen.
* Determine the rate of disease relapse and incidence of post-transplantation lymphoproliferative disease in these patients.

OUTLINE: Patients are stratified according to disease category (malignant vs non-malignant) and graft source (unrelated vs HLA-matched sibling).

Beginning at least 4 weeks after conventional-dose chemotherapy, patients receive non-myeloablative conditioning comprising fludarabine IV over 30 minutes on days -8 to -4, cyclophosphamide IV over 2 hours on days -3 to -2, and anti-thymocyte globulin IV over at least 4 hours on days -2 and -1. Patients undergo filgrastim (G-CSF)-mobilized allogeneic peripheral blood stem cell transplantation on day 0.

Patients are followed weekly for 3 months, every 2 weeks for 3 months, monthly for 6 months, and then every 2 months thereafter.

PROJECTED ACCRUAL: A minimum of 30 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven high-risk hematologic malignancy

  * Acute non-lymphocytic leukemia (ANLL) after induction failure, or in first complete remission (CR) with high-risk features, including any of the following:

    * Stem cell or biphenotypic classification (AML-M0)
    * Erythroleukemia (AML-M6)
    * Acute megakaryocytic leukemia (AML-M7)
    * Cytogenetic markers indicative of poor prognosis
    * Failure to achieve CR after standard induction therapy
  * Acute lymphocytic leukemia (ALL) or ANLL in relapse or second or subsequent remission
  * Chronic myelogenous leukemia (CML) in chronic or accelerated phase

    * Patients with CML in blast crisis are eligible after reinduction chemotherapy places them in chronic phase
  * High-risk ALL in first CR with high risk defined by presence of t(4;11), t(9;22) translocation, hyperleukocytosis (initial WBC greater than 30,000/mm^3), or failure to achieve CR by day 28 after standard induction

    * No T-cell ALL or t(8;14) positive B-cell ALL in first remission with hyperleukocytosis
  * Myelodysplastic syndrome by peripheral blood smear and bone marrow examination

    * Refractory to medical management OR
    * Cytogenetic abnormalities predictive of transformation into acute leukemia including 5q-, 7q-, monosomy 7, and trisomy 8 OR
    * Evidence of evolution to AML (e.g., refractory anemia with excess blasts (RAEB) or RAEB in transformation)
  * Multiple myeloma, non-Hodgkin's lymphoma (NHL), ANLL, or ALL with recurrent disease after autologous stem cell transplantation (SCT)

    * At least 3 months since prior autologous SCT
  * Hodgkin's lymphoma, NHL, or multiple myeloma beyond first CR or primary induction failures whose disease has demonstrated sensitivity to pre-transplantation cytoreduction (defined as greater than 50% reduction in tumor burden)

    * Mantle zone NHL allowed after induction therapy
  * Myeloproliferative disorder that is non-responsive to medical management and requires allografting, unless evidence of grade 3 or worse myelofibrosis on marrow biopsy OR
* Histologically proven acquired severe aplastic anemia (SAA) that is recurrent or unresponsive after anti-thymocyte globulin and/or cyclosporine

  * SAA defined by at least 2 of the following conditions:

    * Granulocyte count less than 500/mm^3
    * Platelet count less than 20,000/mm^3
    * Absolute reticulocyte count less than 20,000/mm^3 after correction for hematocrit
* Ineligible for full ablative conditioning due to any of the following conditions:

  * Prior extensive therapy (more than 2 salvage chemotherapy regimens and/or autologous transplantation)
  * Over age 55 OR
  * Under age 55 with comorbid disease (e.g., suboptimal cardiac, pulmonary, or renal function and/or prior life-threatening infection)
* HLA-A, B, and DR phenotypically identical sibling donor OR
* HLA-A, B, and DR identical genetically matched unrelated donor
* No ANLL in first CR (less than 5% blasts in marrow) with translocations t(8;21) and inv(16) unless failed first-line induction therapy OR
* No ANLL in first CR (less than 5% blasts in marrow) with translocations t(15;17) abnormality unless failed first-line induction therapy OR molecular evidence of persistent disease
* No active CNS disease

PATIENT CHARACTERISTICS:

Age:

* 0 to 70

Performance status:

* Zubrod 0-1
* Karnofsky 80-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* See Disease Characteristics

Hepatic:

* ALT/AST no greater than 4 times normal
* Bilirubin no greater than 2.0 mg/dL

Renal:

* See Disease Characteristics
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* See Disease Characteristics
* Shortening fraction or ejection fraction at least 40% of normal for age by echocardiogram or radionuclide scan
* No clinically significant comorbid illnesses (e.g., myocardial infarction or cerebrovascular accident)

Pulmonary:

* See Disease Characteristics
* FVC and FEV_1 at least 60% of predicted for age
* DLCO at least 60% of predicted for adults

Other:

* No severe neurosensory symptoms (i.e., peripheral neuropathy)
* HIV negative
* Active infection allowed if controlled by appropriate drug therapy
* Not pregnant or nursing
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Recovered from prior therapy
* No concurrent investigational agents unless approved by protocol investigators

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2000-06; Primary Completion 2004-01 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of Donor Engraftment | at 28 days
  Peripheral blood from the donor and patient is obtained for chimerism studies. The primary analysis will consist of estimating the graft failure proportions for each of the separate patient groups and calculating confidence intervals for these proportions. This analysis will be done conditional on patients surviving at least 28 days.

SECONDARY OUTCOMES:
Stable donor hematopoietic chimerism | at day 100
  Number of Patients Transplanted More Than 100 Days Ago
Event free and overall survival | to progression/death

CONTACTS AND LOCATIONS:
Overall Officials: Tamila Kindwall-Keller, DO, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States